CLINICAL TRIAL: NCT04759027
Title: Prospective Evaluation of the Reliability and Re-applicability of Subacromial Distance Measurement With Standard Radiographic Imaging Compared to Ultrasound Imaging
Brief Title: Reliability of the Subacromial Distance Measurements With Standard Radiographic Imaging
Status: Completed | Type: Observational
Sponsor: Göker Utku değer (Other)
Responsible Party: Sponsor-Investigator, Göker Utku değer, Research assistant, Istanbul University - Cerrahpasa
Organization: Istanbul University - Cerrahpasa (Other)
Other Study IDs: E-83045809-604.01.02-1214
Record Dates: First submitted 2021-02-01; First posted 2021-02-17 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Subacromial Impingement; Rotator Cuff Tears
Keywords: x-ray; direct radiography; ultrasound; acromiohumeral distance; subacromial distance; rotator cuff
MeSH Terms: conditions — Shoulder Impingement Syndrome; Rotator Cuff Injuries

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- X-ray: Measurements of subacromial distance on standardized direct radiography
  Interventions: Other: subacromial distance measurement
- ultrasound: Measurements of subacromial distance on ultrasound
  Interventions: Other: subacromial distance measurement

INTERVENTIONS:
Other: subacromial distance measurement — distance between acromion and humerus

SUMMARY:
Patients with complaints of shoulder pain or limitation of motion, who admitted to outpatient orthopaedic clinic will be analyzed. It was planned to measure the subacromial distance using standardized both shoulder ap, true ap and outlet radiographs, and ultrasound to be performed for shoulder circumference soft tissue and muscle-tendon evaluation. The measurement made by the physical therapy and rehabilitation specialist with ultrasound will be considered to be accurate, and it was planned to evaluate the reliability of the graphy measurements by comparing this measurement with the measurements in the graphs. In addition, it was planned to evaluate the intra-observer and inter-observer compliance by re-measuring the subacromial distance on the radiograph by orthopedic doctors of three different seniority levels with an interval of one month.

DETAILED DESCRIPTION:
Rotator cuff injuries are the most common injury to the shoulder girdle. Patients present to the clinic with shoulder compression at an early age and with tears in older ages. Nearly 50% of the population can be torn in advanced ages. Repetitive trauma caused by overuse is blamed for rotator cuff tears. The narrowing of the subacromial distance causes compression in the anterior, tears and enlargement of the tears by extrinsic mechanism. In addition, the surgery to be performed according to the subacromial distance and the benefit to the patient from this surgery can be predicted. In studies conducted in normal population, subacromial distance was reported to be between 6-12 mm, measurements made under 6-7 mm were evaluated as pathologically and were defined as tears that would not benefit from repair.

The reliability of this measurement, which guides the diagnosis and treatment, is important. The diagnosis of these diseases is made by imaging methods following the physical examination and then the decision of the appropriate treatment method is made. It is known that conventional radiographs constitute the first step of evaluation as a standard in almost all patients in orthopedic practice. Magnetic resonance imaging and ultrasound are often preferred for shoulder, shoulder circumference pathology and injuries, in relation to the examination findings after direct radiography at the diagnosis and examination stage. Drawing graphs on both shoulders from these images to provide comparative evaluation provides more detailed information in evaluation. The subacromial distance or acromiohumeral distance used in the evaluation of rotator cuff pathologies was defined as the shortest distance between the sclerotic inferior border of the acromion and the humeral head. The measurement of this distance can be made with direct graphy, mri, ct, and ultrasound. In the only systematic review on this subject, it was emphasized that this measurement can be made with ultrasound as the most reliable, and the evaluations made by direct radiography are worthless. In these inferences, the poor methodology of the studies made using direct graphy measurement was shown as the reason. Many studies have been carried out by standardizing the imaging, its importance has been proven by the inconsistent results of the study with non-standardized graphs.

ELIGIBILITY:
Inclusion Criteria:

* shoulder pain ( acute traumatic or non-traumatic chronic)

Exclusion Criteria:

* end stage glenohumeral joint arthrosis
* adhesive capsulitis
* fractures
* previous shoulder surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients over the age of 18 who admitted to orthopedics and traumatology outpatient clinics with a complaint of non-traumatic shoulder pain for more than two weeks or traumatic shoulder pain will be study population.
Sampling Method: Non-Probability Sample
Enrollment: 56 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
RELIABILITY OF DIRECT RADIOGRAPHY IMAGING | within 2 weeks after first evaluation
  The investigators will compare the results of subacromial distance measure on X-ray and ultrasound. Ultrasound measures were accepted as gold standart method.

SECONDARY OUTCOMES:
REPRODUCIBLITY | 1 month apart measurements will be evaluate
  if X-ray measurements will correlate with ultrasound, the investigators will evaluate intraobserver and interobserver measurement differences

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet F Guven, Assoc.prof, Study Director — Istanbul University-Cerrahpasa, Cerrahpasa Medical Faculty
Locations (1):
- Istanbul University- Cerrahpasa Cerrahpasa Medical Faculty, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Luime JJ, Koes BW, Hendriksen IJ, Burdorf A, Verhagen AP, Miedema HS, Verhaar JA. Prevalence and incidence of shoulder pain in the general population; a systematic review. Scand J Rheumatol. 2004;33(2):73-81. doi: 10.1080/03009740310004667. PMID 15163107
- [Background] Tempelhof S, Rupp S, Seil R. Age-related prevalence of rotator cuff tears in asymptomatic shoulders. J Shoulder Elbow Surg. 1999 Jul-Aug;8(4):296-9. doi: 10.1016/s1058-2746(99)90148-9. PMID 10471998
- [Background] Yamamoto A, Takagishi K, Osawa T, Yanagawa T, Nakajima D, Shitara H, Kobayashi T. Prevalence and risk factors of a rotator cuff tear in the general population. J Shoulder Elbow Surg. 2010 Jan;19(1):116-20. doi: 10.1016/j.jse.2009.04.006. PMID 19540777
- [Background] Azzoni R, Cabitza P, Parrini M. Sonographic evaluation of subacromial space. Ultrasonics. 2004 Apr;42(1-9):683-7. doi: 10.1016/j.ultras.2003.11.015. PMID 15047367
- [Background] Saupe N, Pfirrmann CW, Schmid MR, Jost B, Werner CM, Zanetti M. Association between rotator cuff abnormalities and reduced acromiohumeral distance. AJR Am J Roentgenol. 2006 Aug;187(2):376-82. doi: 10.2214/AJR.05.0435. PMID 16861541
- [Background] Schmidt WA, Schmidt H, Schicke B, Gromnica-Ihle E. Standard reference values for musculoskeletal ultrasonography. Ann Rheum Dis. 2004 Aug;63(8):988-94. doi: 10.1136/ard.2003.015081. PMID 15249327
- [Background] Norwood LA, Barrack R, Jacobson KE. Clinical presentation of complete tears of the rotator cuff. J Bone Joint Surg Am. 1989 Apr;71(4):499-505. PMID 2703509
- [Background] Ellman H, Hanker G, Bayer M. Repair of the rotator cuff. End-result study of factors influencing reconstruction. J Bone Joint Surg Am. 1986 Oct;68(8):1136-44. PMID 3771595
- [Background] Kum DH, Kim JH, Park KM, Lee ES, Park YB, Yoo JC. Acromion Index in Korean Population and Its Relationship with Rotator Cuff Tears. Clin Orthop Surg. 2017 Jun;9(2):218-222. doi: 10.4055/cios.2017.9.2.218. Epub 2017 May 8. PMID 28567226
- [Background] Mayerhoefer ME, Breitenseher MJ, Wurnig C, Roposch A. Shoulder impingement: relationship of clinical symptoms and imaging criteria. Clin J Sport Med. 2009 Mar;19(2):83-9. doi: 10.1097/JSM.0b013e318198e2e3. PMID 19451760
- [Background] Werner CM, Conrad SJ, Meyer DC, Keller A, Hodler J, Gerber C. Intermethod agreement and interobserver correlation of radiologic acromiohumeral distance measurements. J Shoulder Elbow Surg. 2008 Mar-Apr;17(2):237-40. doi: 10.1016/j.jse.2007.06.002. Epub 2007 Dec 26. PMID 18162412
- [Background] Sasiponganan C, Dessouky R, Ashikyan O, Pezeshk P, McCrum C, Xi Y, Chhabra A. Subacromial impingement anatomy and its association with rotator cuff pathology in women: radiograph and MRI correlation, a retrospective evaluation. Skeletal Radiol. 2019 May;48(5):781-790. doi: 10.1007/s00256-018-3096-0. Epub 2018 Oct 27. PMID 30368566
- [Background] Yoshida Y, Matsumura N, Yamada Y, Yamada M, Yokoyama Y, Matsumoto M, Nakamura M, Nagura T, Jinzaki M. Evaluation of three-dimensional acromiohumeral distance in the standing position and comparison with its conventional measuring methods. J Orthop Surg Res. 2020 Sep 23;15(1):436. doi: 10.1186/s13018-020-01935-9. PMID 32967710
- [Background] van de Sande MA, Rozing PM. Proximal migration can be measured accurately on standardized anteroposterior shoulder radiographs. Clin Orthop Relat Res. 2006 Feb;443:260-5. doi: 10.1097/01.blo.0000196043.34789.73. PMID 16462449
- [Background] Ueda Y, Tanaka H, Tomita K, Tachibana T, Inui H, Nobuhara K, Umehara J, Ichihashi N. Comparison of shoulder muscle strength, cross-sectional area, acromiohumeral distance, and thickness of the supraspinatus tendon between symptomatic and asymptomatic patients with rotator cuff tears. J Shoulder Elbow Surg. 2020 Oct;29(10):2043-2050. doi: 10.1016/j.jse.2020.02.017. Epub 2020 May 26. PMID 32471753
- [Background] Xu M, Li Z, Zhou Y, Ji B, Tian S, Chen G. Correlation between acromiohumeral distance and the severity of supraspinatus tendon tear by ultrasound imaging in a Chinese population. BMC Musculoskelet Disord. 2020 Feb 17;21(1):106. doi: 10.1186/s12891-020-3109-8. PMID 32066419
- [Background] Pijls BG, Kok FP, Penning LI, Guldemond NA, Arens HJ. Reliability study of the sonographic measurement of the acromiohumeral distance in symptomatic patients. J Clin Ultrasound. 2010 Mar-Apr;38(3):128-34. doi: 10.1002/jcu.20674. PMID 20127966
- [Background] McCreesh KM, Crotty JM, Lewis JS. Acromiohumeral distance measurement in rotator cuff tendinopathy: is there a reliable, clinically applicable method? A systematic review. Br J Sports Med. 2015 Mar;49(5):298-305. doi: 10.1136/bjsports-2012-092063. Epub 2013 Jul 2. PMID 25690908
- [Background] Fehringer EV, Rosipal CE, Rhodes DA, Lauder AJ, Puumala SE, Feschuk CA, Mormino MA, Hartigan DE. The radiographic acromiohumeral interval is affected by arm and radiographic beam position. Skeletal Radiol. 2008 Jun;37(6):535-9. doi: 10.1007/s00256-008-0467-y. PMID 18343920